CLINICAL TRIAL: NCT01642199
Title: A Randomized Trial Testing Lay Health Coaches for Obesity Treatment
Brief Title: Lay Health Coaches for Weight Loss: Peers Versus Mentors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Tricia Leahey, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01DK095771-01 (NIH)
Record Dates: First submitted 2012-07-12; First posted 2012-07-17 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Obesity
Keywords: obesity; weight loss; lay health coach; peer coach; mentor coach; reduced intensity weight loss program
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Reduced Intensity Behavioral Weight Loss + Peer Health Coach (Active Comparator)
  Interventions: Behavioral: Reduced Intensity Behavioral Weight Loss + Peer Health Coach
- Reduced Intensity Behavioral Weight Loss + Mentor Health Coach (Active Comparator)
  Interventions: Behavioral: Reduced Intensity Behavioral Weight Loss + Mentor Health Coach
- Reduced Intensity Behavioral Weight Loss (Active Comparator)
  Interventions: Behavioral: Reduced Intensity Behavioral Weight Loss

INTERVENTIONS:
Behavioral: Reduced Intensity Behavioral Weight Loss + Peer Health Coach — Participants will receive a 12-month reduced intensity group behavioral weight loss program. During weeks that there are no group meetings, participants will be coached by peers (i.e., other members of their weight loss group).
  Arms: Reduced Intensity Behavioral Weight Loss + Peer Health Coach
Behavioral: Reduced Intensity Behavioral Weight Loss + Mentor Health Coach — Participants will receive a 12-month reduced intensity group behavioral weight loss program. During weeks that there are no group meetings, participants will be coached by a mentor (i.e., successful weight loser).
  Arms: Reduced Intensity Behavioral Weight Loss + Mentor Health Coach
Behavioral: Reduced Intensity Behavioral Weight Loss — Participants will receive 12 months of a reduced intensity group behavioral weight loss program.
  Arms: Reduced Intensity Behavioral Weight Loss

SUMMARY:
The primary aim of this study is to determine whether reduced intensity behavioral weight loss treatment (rBWL) + Peer Health Coaches yields significantly greater weight loss than rBWL + Mentor Health Coaches and rBWL alone.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 30 and 40
* Age between 40 and 60 years
* English speaking

Exclusion Criteria:

* Are unwilling to communicate regularly with a weight loss coach
* Report not being able to walk 2 blocks (1/4 mile) without stopping
* Are currently participating in a weight loss program, taking a weight loss medication, have a history of bariatric surgery, or lost ≥ 5% of body weight during the past 6-months
* Are pregnant, lactating, less than 6-months post-partum, or plan to become pregnant during the intervention timeframe
* Report a heart condition, chest pain during periods of rest or activity, or loss of consciousness on the Physical Activity Readiness Questionnaire
* Report a medical condition that would jeopardize their safety if involved in a weight management program with diet and exercise guidelines
* Report conditions that, in the judgment of the PI, would render the participant unlikely to follow the study protocol (e.g., relocation, dementia, terminal illness, substance abuse).

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 278 (Actual)
Dates: Start 2013-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Weight change from the initial assessment to the 12-month assessment measured on a digital scale to the nearest 0.1-kilogram | baseline to 12 months

SECONDARY OUTCOMES:
Direction of social comparison between participants and their Peer or Mentor weight loss coach | 2-weeks, 3-months, 6-months, 9-months, and 12-months
  Participants in rBWL + Peer and rBWL + Mentor will complete a questionnaire that assesses whether their progress on weight loss, diet, and activity are "worse," "similar to," or "better" than their coach's on a 5-point likert scale. Mean scores on this measure will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Tricia M Leahey, PhD, Principal Investigator — The Miriam Hospital / Warren Alpert Medical School at Brown University
Locations (1):
- The Miriam Hospital's Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Leahey TM, Huedo-Medina TB, Grenga A, Gay L, Fernandes D, Denmat Z, Doyle C, Areny-Joval R, Wing RR. Patient-provided e-support in reduced intensity obesity treatment: The INSPIRE randomized controlled trial. Health Psychol. 2020 Dec;39(12):1037-1047. doi: 10.1037/hea0000996. PMID 33252929